CLINICAL TRIAL: NCT06969482
Title: The Effect of Patient Advocacy Training on Advocacy Skills, Ethical Sensitivity and Patient Safety Culture in Nurses: A Randomized Controlled Study
Brief Title: The Effect of Patient Advocacy Training on Advocacy Skills, Ethical Sensitivity, and Patient Safety Culture in Nurses
Acronym: (RCT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Neslihan Şahin, Doctoral Student, Selcuk University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 203172001002
Record Dates: First submitted 2025-03-18; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Education
Keywords: Patient Advocacy, Ethics, Patient Safety
MeSH Terms: interventions — Early Intervention, Educational; Randomized Controlled Trials as Topic

STUDY DESIGN:
Intervention Model Description: Control and intervention group nurses will receive routine training provided by the Hospital Education and Quality Unit. After obtaining informed consent and conducting pre-tests, the 70 nurses forming the study group will be randomly assigned to the experimental and control groups using simple randomization. Subsequently, the intervention group of 35 nurses will receive 8 weeks of training. After the training, both groups will undergo post-tests.
  The tools used for evaluation are as follows:
  * Personal Information Form
  * Patient Advocacy Scale for Nurses
  * Moral Sensitivity Questionnaire
  * Patient Safety Culture Hospital Questionnaire
  These tools will be administered and evaluated by a specialist nurse in both groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effect of Patient Advocacy Training on Advocacy Skills, Ethical Sensitivity and Patient Safety C (No Intervention): In this application, measurements are made before the experiment/intervention (pre-test).
- Pre-testing was applied to all individuals participating in the study. (Active Comparator): Post-training measurements of the experimental group and pre-test and post-test comparison analyses of the two groups.
  Interventions: Behavioral: measuring knowledge level; Other: educational intervention

INTERVENTIONS:
Behavioral: measuring knowledge level — The study group consists of 70 nurses, each consisting of 35 people. After the routine training of the hospital was given to the control and experimental groups, their consents were obtained and the pre-tests were completed, they were divided into experimental and control groups using simple randomization. The first group of nurses in the control group will not receive any intervention other than the routine training given by the hospital.
  Arms: Pre-testing was applied to all individuals participating in the study.
Other: educational intervention — the effectiveness of training by making measurements after training and comparing them with pre-training results
  Other Names: randomized controlled trial
  Arms: Pre-testing was applied to all individuals participating in the study.

SUMMARY:
In this study, the aim is to evaluate the effects of patient advocacy training provided to nurses on their advocacy skills, ethical sensitivity, and patient safety culture level.

DETAILED DESCRIPTION:
This research is a Randomized Controlled Trial (RCT) conducted to investigate the impact of patient advocacy training on nurses by evaluating its effectiveness in increasing nurses' ethical sensitivity and promoting a positive patient safety culture through Bloom's Taxonomy. This study, which will deeply examine the relationship between patient advocacy training, ethical sensitivity, and patient safety culture, aims to provide evidence-based insights that can inform nursing education, training programs, and healthcare policies, ultimately contributing to the improvement of patient outcomes and the overall quality of healthcare delivery.

ELIGIBILITY:
Inclusion Criteria: Employees who have no obstacles to participating in the training program Exclusion Criteria: Having worked in the hospital for at least six months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-21 (Estimated); Primary Completion 2025-07-27 (Estimated); Study Completion 2025-09-19 (Estimated)

PRIMARY OUTCOMES:
Patient advocacy scale, Moral sensitivity survey, Patient Safety Culture Hospital Survey | up to 8 weeks
  Patient advocacy scale total and sub-dimension scores Moral Sensitivity Questionnaire scale total and sub-dimension scores Evaluation of Patient Safety Culture Hospital Survey is Made Only Based on Positive Response Average Scores
Patient Advocacy Scale for Nurses, Moral Sensitivity Questionnaire (ADA),Hospital Patient Safety Culture Survey (HSOPSC) | up to 8 weeks
  Patient Advocacy Scale for Nurses (HSO) Consists of 39 items and 7 sub-dimensions.- Scoring: Total score ranges from 39 to 195; higher scores indicate higher level of advocacy
  * Reliability: Cronbach alpha coefficient 0.95; ranges from 0.82 to 0.92 for sub-dimensions Moral Sensitivity Questionnaire (ADA) Consists of 30 items and 6 sub-dimensions,- Scoring: Total score ranges from 30 to 210; lower scores indicate higher ethical sensitivity
  * Reliability: Cronbach alpha coefficient ranges from 0.82 to 0.84; test-retest correlation coefficient ranges from 0.81 to 0.99 Patient Safety Culture Survey (HSOPSC)
  * Contains a total of 42 items, assesses patient safety culture in 12 dimensions, Scoring: Each item is assessed using a 5-point Likert scale (1=Strongly disagree, 5=Strongly agree) Reliability: Validity and reliability studies of the Turkish version have been conducted

SECONDARY OUTCOMES:
Educational intervention | after 8 weeks
  Patient Advocacy Scale for Nurses (HSO) Consists of 39 items and 7 sub-dimensions.- Scoring: Total score ranges from 39 to 195; higher scores indicate higher level of advocacy
  * Reliability: Cronbach alpha coefficient 0.95; ranges from 0.82 to 0.92 for sub-dimensions Moral Sensitivity Questionnaire (ADA) Consists of 30 items and 6 sub-dimensions,- Scoring: Total score ranges from 30 to 210; lower scores indicate higher ethical sensitivity
  * Reliability: Cronbach alpha coefficient ranges from 0.82 to 0.84; test-retest correlation coefficient ranges from 0.81 to 0.99 Patient Safety Culture Survey (HSOPSC)
  * Contains a total of 42 items, assesses patient safety culture in 12 dimensions, Scoring: Each item is assessed using a 5-point Likert scale (1=Strongly disagree, 5=Strongly agree) Reliability: Validity and reliability studies of the Turkish version have been conducted
Post-tests after 8 weeks of training | 1 month
  Pre-tests of Both Groups Comparison of Experimental Group According to Follow-up Times Post-tests of Both Groups Should Also Be Done and Reported

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Ş Doctoral student, Doctoral student, Principal Investigator — Selcuk University; Neslihan Ş ŞAHİN, Doctoral student, Principal Investigator — Selcuk University

IPD SHARING:
Plan to Share IPD: No